CLINICAL TRIAL: NCT06616857
Title: Personalized Mobile Health Platform to Promote Physical Activity in Adolescents and Young Adults With Cystic Fibrosis
Acronym: NUDGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, David Fedele, Principal Research Scientist, Nemours Children's Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2158063; 003780A122 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2024-09-20; First posted 2024-09-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis (CF)
Keywords: physical activity
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NUDGE (Experimental)
  Interventions: Behavioral: NUDGE
- Education (Active Comparator)
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: NUDGE — Individuals in this condition will receive intervention content to promote physical activity.
  Arms: NUDGE
Other: Education — Individuals will receive educational materials about how to increase physical activity
  Arms: Education

SUMMARY:
The goal of this clinical trial is to help adolescents and young adults between the ages of 13-25 with Cystic Fibrosis (CF), medically stable, able to speak and read English, and are not experiencing a CF - related exacerbation, who are already active to remain, or gradually encourage them to increase their levels of physical activity

Participants will be asked to utilize a smartphone program, called NUDGE that we have developed. NUDGE is a chatbot with evidence-based features known to help teens make progress toward health goal:

* Set and review goals
* Self-monitor progress
* Provide feedback on goal attainment
* Revise future goals

DETAILED DESCRIPTION:
The goal of this study is to conduct a 6-month delayed treatment pilot Trial with adolescents and young adults (AYA) ages 13-25 with Cystic Fibrosis (CF) or a CF related disorder) to establish feasibility and obtain data necessary to inform a Phase III efficacy trial. AYAs 18 years-old and caregivers of AYAs 13-17 years-old will complete the informed consent process. AYAs 13-17 years-old will be asked to assent to participate in the study. After completion of the baseline study measures and return of actigraphy monitors, staff will notify AYAs of their randomized assignment. AYAs receiving NUDGE will then begin receiving intervention content for 6 months. AYAs randomized to control will receive NUDGE at the conclusion of the Month 3 study visit. Study visits will occur at Months 0, 3, and 6 with staff masked to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

1. 13-25 years old
2. Has a verified CF diagnosis or CF-related disorder
3. Medically stable (i.e., FEV1>30%, not experiencing a CF-related exacerbation)
4. Speaks and reads English

Exclusion Criteria:

1. Have a comorbidity limiting PA participation (e.g., neurological condition)
2. Have a significant cognitive impairment that interferes with study completion
3. Have any oxygen, CPAP or BiPAP requirement

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Baseline
  Recruitment: Our recruitment goal is 30 AYAs with CF.
Retention | 3-month
  Retention: Our criterion for success is no more than 20% attrition.
Engagement | 3-month
  Engagement: We will be considered engagement a success if AYAs in NUDGE respond to an average of 4/7 (57%) messages each week during the first 3 months that a participant uses NUDGE.
Acceptability | 3-month
  Acceptability: We will consider NUDGE acceptable if users report a satisfaction rating of ≥3 (mostly satisfied) on our modified Client Satisfaction Questionnaire and rate it as usable as ≥70% of other computerized systems on the System Usability Scale. We will also be attentive to themes in relation to the barriers and facilitators of using NUDGE and its success in promoting PA in interviews.

SECONDARY OUTCOMES:
Actigraphy | Baseline, 3-month, and 6-month
  We will objectively measure AYA's moderate-to-vigorous PA for 7-days via ActiGraph wGT3X-BT accelerometers. All data will be processed using Actilife software. We will remove periods of non-wear and sleep; days with >10-hours of valid data during waking hours will be retained. Data will be binned into 15 second epochs and processed using the Chandler algorithm.
Lung Functioning | Baseline, 3-month, and 6-month
  Lung function will be assessed for 7-days via the AM1+ portable spirometer. AYAs will undergo a standardize training and complete three maximal effort blows every morning and evening. The main outcomes will be forced expiratory volume in one second (FEV1) percent predicted.
CF Quality of Life | Baseline, 3-month, and 6-month
  AYA CF-related quality of life will be assessed via the Cystic Fibrosis Questionnaire-Revised.

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Childrens Health, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plans to share IPD will need to be discussed with the IRB.